CLINICAL TRIAL: NCT06857630
Title: The Association Between Preoperative Hemoglobin and Acute Kidney Injury in Emergency Surgery: A Prospective Observational Study
Brief Title: Preoperative Hemoglobin and Acute Kidney Injury in Emergency Surgery
Status: Recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2024/19/4
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Emergency Surgery; Acute Kidney Injury; Hemoglobin
Keywords: Acute kidney injury; Emergency surgery; Risk factor; Hemoglobin
MeSH Terms: conditions — Acute Kidney Injury | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group AKI: Postoperative renal failure
  Interventions: Other: Observational
- Group non-AKI: Postoperative non renal failure
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Postoperative acute kidney injury and hemoglobin level relationship observation

SUMMARY:
Optimization of hemoglobin levels for organ perfusion is essential, especially in critically ill patients. Although anemia is associated with severe organ failure, especially in coronary artery disease, the effects of blood transfusion or various interventions to increase hemoglobin levels on outcomes continue to be debated. The effects of hemoglobin levels in emergency surgery patients on the development of postoperative AKI have been investigated in a small number of studies in the literature, and clear results have not yet been reported. This study was designed to evaluate the effect of hemoglobin levels on the development of AKI after adjustment for known predictive factors.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication in patients undergoing major surgery and is associated with both short-term morbidity and mortality and long-term adverse outcomes including the development of Chronic Kidney Failure. Optimization of hemoglobin levels for organ perfusion is essential, especially in critically ill patients. Although anemia is associated with severe organ failure, especially in coronary artery disease, the effects of various interventions such as blood transfusion or increasing hemoglobin levels on outcomes continue to be debated. This prospective observational study was planned to evaluate the effect of hemoglobin levels before emergency surgery on the development of postoperative AKI.

Emergency operated patients will be divided into two groups as Group AKI and Group non-AKI according to the development of postoperative renal failure. Postoperative AKI diagnosis and severity will be evaluated according to serum creatinine and/or urine output according to KDIGO (Kidney Disease: Improving Global Outcomes criteria).

Demographic characteristics of the patients, preoperative complete blood count, blood biochemistry characteristics, hemodynamic variables, fluid replacement, blood and blood product replacements, surgical characteristics, development and severity of AKI in the postoperative period will be recorded and the effect of hemoglobin level on the development of AKI will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergency non-cardiac surgery

Exclusion Criteria:

* Known renal failure
* Need for reoperation within 48 hours postoperatively
* Exit status within 48 hours postoperatively
* Known hematological disease
* Known kidney transplantation
* Urgent surgery planned due to urinary system related diseases
* Patients who did not accept to participate in the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing emergency non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Acute renal failure. | 72 hours
  The effect of hemoglobin level before emergency surgery on the development of postoperative acute renal failure.

SECONDARY OUTCOMES:
Hospital days | 1 month
  The effect of hemoglobin level before emergency surgery on the hospital days

CONTACTS AND LOCATIONS:
Overall Officials: özgür kömürcü, 1, Study Director — Samsun University
Locations (1):
- Özgür Kömürcü, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meersch M, Schmidt C, Zarbock A. Perioperative Acute Kidney Injury: An Under-Recognized Problem. Anesth Analg. 2017 Oct;125(4):1223-1232. doi: 10.1213/ANE.0000000000002369. PMID 28787339
- [Background] Grams ME, Sang Y, Coresh J, Ballew S, Matsushita K, Molnar MZ, Szabo Z, Kalantar-Zadeh K, Kovesdy CP. Acute Kidney Injury After Major Surgery: A Retrospective Analysis of Veterans Health Administration Data. Am J Kidney Dis. 2016 Jun;67(6):872-80. doi: 10.1053/j.ajkd.2015.07.022. Epub 2015 Sep 1. PMID 26337133
- [Background] Cabezuelo JB, Ramirez P, Rios A, Acosta F, Torres D, Sansano T, Pons JA, Bru M, Montoya M, Bueno FS, Robles R, Parrilla P. Risk factors of acute renal failure after liver transplantation. Kidney Int. 2006 Mar;69(6):1073-80. doi: 10.1038/sj.ki.5000216. PMID 16528257